CLINICAL TRIAL: NCT05500066
Title: AEQUALIS™ FLEX REVIVE™ Study (REVIVE)
Acronym: REVIVE
Status: Enrolling by invitation | Type: Observational
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: 20F-W-REVIVE-RM
Record Dates: First submitted 2022-08-04; First posted 2022-08-12 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis Shoulder; Fractures Humerus; Avascular Necrosis; Correction of Functional Deformity; Traumatic Arthritis; Revision of Other Devices if Sufficient Bone Stock Remains; Rotator Cuff Tears
Keywords: Total Shoulder Replacement; Osteoarthritis; Joint Diseases; Musculoskeletal Diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Humeral Fractures; Osteonecrosis; Rotator Cuff Injuries; Osteoarthritis; Joint Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Aequalis Flex Revive Shoulder System: Commercially available shoulder system available in both anatomic and reversed configurations.
  Interventions: Device: Aequalis Flex Revive Shoulder System

INTERVENTIONS:
Device: Aequalis Flex Revive Shoulder System — The AEQUALIS FLEX REVIVE Shoulder System is intended for use as:
  * A replacement of shoulder joints in primary anatomic or in primary reverse
  * A replacement of other shoulder joints devices in case of revisions if sufficient bone stock remains.
  The system also allows for conversion from anatomic to reverse shoulder prosthesis in case of revision.

SUMMARY:
This is an international, single arm, multicenter, prospective, non-significant risk, Post-Market Clinical Follow-up (PMCF) study. Data will be collected for the commercially available AEQUALIS FLEX REVIVE shoulder system in both the anatomic and reversed configurations.

The purpose of this study is to collect data needed to satisfy the European Union (EU) Medical Device Regulation (MDR) clinical post-market surveillance (PMS) and reporting requirements, and to support future regulatory submissions and peer-reviewed publications on device performance and safety.

DETAILED DESCRIPTION:
This is an international, single arm, multicenter, prospective, non-significant risk, Post-Market Clinical Follow-up (PMCF) study. Data will be collected for the commercially available AEQUALIS FLEX REVIVE shoulder system in both the anatomic and reversed configurations.

The primary outcome measure will be measured by the average improvement in American Shoulder and Elbow Surgeons (ASES) score from baseline to 24 months.

Secondary outcome measures include patient reported outcome measures (PROMs) and standard radiographic findings, including, but not limited to: device migration, component breakage, and bone characteristics.

Device revision and adverse events (AEs) will be assessed annually throughout the study. Range of motion and radiographic imaging assessments will also be performed at Years 1, 2, 5 and 10 post-operation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of the informed consent.
* Informed and willing to sign an informed consent form approved by IRB or Ethics Committee (EC) (when applicable).
* Willing and able to comply with the requirements of the study protocol.
* Considered for a candidate for shoulder arthroplasty using the study device
* Meets indications for use requirements or other local, regional, or geographic specific regulatory requirements

Exclusion Criteria:

* Not able to comply with the study procedures based on the judgment of the assessor (e.g., cannot comprehend study questions, inability to keep scheduled assessment times)
* Patient belongs to a vulnerable group of patients, including minor patients, those unable to decide for themselves to participate or needing a Legally Authorized Representative (LAR), or others who could be subject to coercion (patients who may not be acting on their own initiative) (referred as "vulnerable subject" in the section 3.44 of the ISO 14155 norm).
* Active local or systemic infection, sepsis, or osteomyelitis
* Poor bone quality, where there could be considerable migration of the prothesis and/or a chance of fracture of the humerus or glenoid (reassessed at time of surgery)
* Significant injury to the brachial plexus
* Inadequate bone stock in the proximal humerus or glenoid fossa for supporting the components
* Neuromuscular disease (e.g., joint neuropathy)
* Patient with known allergy to one of the product materials
* Metabolic disorders which may impair bone formation
* Patient pregnancy
* Planned for two-stage surgery (reassessed at time of surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 110 subjects are to be enrolled in this clinical investigation. Subjects participating in this clinical investigation will be recruited from the investigator's standard subject population, where all subjects presenting for an anatomic or reversed total shoulder arthroplasty will be evaluated for clinical investigation participation based on the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2028-01-06 (Estimated); Study Completion 2036-01-03 (Estimated)

PRIMARY OUTCOMES:
Average Improvement from Baseline to last follow-up visit in ASES Score | 24 Month
  ASES Score = American Shoulder and Elbow Surgeons Score, 11 items with total score reported out of 100 measuring pain and activity of patient's evaluated shoulder where lower scores indicate more pain and less function

SECONDARY OUTCOMES:
Constant Score | through study completion, an average of 1 year
  A score based on a 100-point scale determined by objective measurements made by the physician in the clinic and subjective values based on pain and activities of daily living reported by the patient.
SANE | through study completion, an average of 1 year
  Single question that asks the patient to rate their shoulder on a scale from 0 to 100, where 100 is normal.
EQ 5-D | through study completion, an average of 1 year
  Consists of a 5-question measure where patients rate their health today on a 5-point scale on a 5-dimension scale and a visual analogue scale to measure overall health status.
Patient Satisfaction | through study completion, an average of 1 year
  Single subjective question "How satisfied are you with your shoulder?"
Radiographic Findings | Baseline, 1 year, 2 year, 5 year and 10 year
  Images will be reviewed by a single orthopedic surgeon to assess for standard radiographic findings, including, but not limited to: device migration, component breakage, and bone characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur de Gast, MD MSc PhD, Study Director — Stryker Trauma and Extremities
Locations (4):
- United States (4):
  - Western Orthopaedics, P.C., Denver, Colorado
  - Coastal Orthopedics, Bradenton, Florida
  - Foundation for Orthopaedic Research & Education, Tampa, Florida
  - Baptist Health Lexington, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: No